CLINICAL TRIAL: NCT01105000
Title: The Role of Socioeconomic Status and Ethnicity in Influencing HPV Vaccine Knowledge and Attitudes in Adult Women
Brief Title: Human Papilloma Virus (HPV) Knowledge and Attitudes and the Role of (SES) Socioeconomic Status and Ethnicity
Status: Completed | Type: Observational
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 08-326
Record Dates: First submitted 2010-04-14; First posted 2010-04-16 (Estimated); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: HPV
Keywords: HPV; HPV vaccine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a survey study to assess the vaccination knowledge and attitudes of women in an inner city Gynecology clinic. Results of this study will help determine which factors influence vaccination knowledge and attitudes. This may help improve future vaccination tools.

ELIGIBILITY:
Inclusion Criteria:

* all women attending gynecology clinic

Exclusion Criteria:

* none

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Women attending Gynecology clinic
Sampling Method: Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2008-09; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)